CLINICAL TRIAL: NCT01987310
Title: Assessment of Endothelial Function in Patients With Non Alcoholic Fatty Liver Disease and the Impact of Statin Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was stopped because of lack of interest
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ziv Ben-Ari MD, Head of Disease Medical Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0694-ZBE-CTIL
Record Dates: First submitted 2013-10-27; First posted 2013-11-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; endothelial function; liver steatosis; liver fibrosis; statin treatment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Statin (Active Comparator): statin therapy (atorvastatin 20 mg/d) for 6 months
  Interventions: Drug: atorvastatin
- usual care (No Intervention): follow up group with no intervention
- lifestyle counseling (Active Comparator): lifestyle modification by dietician counseling and follow-up
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 20 mg per day for 6 months
  Other Names: Atorvastatin Teva, Lipitor, Litorva
  Arms: Statin
Behavioral: lifestyle counseling — lifestyle modification by dietician counseling and follow up
  Arms: lifestyle counseling

SUMMARY:
The aim of the current study is to evaluate the association of fatty liver severity and endothelial function in Non-Alcoholic Fatty Liver Disease (NAFLD) patients and to find the impact of statin treatment compared to usual care or life style modification on endothelial function, liver steatosis and fibrosis.

DETAILED DESCRIPTION:
The study cohort will include 150 patients with fatty liver per ultrasound or histology. The patients will be divided randomly to one of three arms: follow up group, lifestyle modification group, and statins therapy (Atorvastatin 20mg/d for 6 months). at screening, after 6 months (end of treatment), and 12 months the patients will undergo:

1. complete physical examination
2. blood pressure measurement
3. assessment of height and weight, body mass index and waist circumference
4. blood samples for complete blood count, fasting plasma glucose, fasting plasma insulin, lipid profile, liver enzymes, albumin, bilirubin, Prothrombin time (PT INR), Hemoglobin A1c, ferritin, adiponectin, C-reactive protein, Tumor necrosis factor alpha, Lipoprotein-phospholipase A2, Apolipoproteins B100, A1, C3, C4, ceruloplasmin
5. Liver elastography and sonographic liver fat quantification
6. Brachial artery flow-mediated dilatation (FMD) measurement

ELIGIBILITY:
Inclusion Criteria:

* subjects willing to comply with study requirements and have signed an informed consent form
* fatty liver per abdominal ultrasound or liver biopsy

Exclusion Criteria:

* alcohol drinking >140g/week
* presence of hepatitis B or C or HIV
* known liver disease other than fatty liver
* usage of drugs known to cause liver steatosis
* subjects with known allergies or hypersensitivity to statins
* subjects with known cardiovascular/cerebrovascular disease
* subjects with known dyslipidemia requiring drug treatment
* subjects with diabetes mellitus
* history of drug or alcohol abuse
* refusal to sig the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in liver steatosis at 6 months | baseline, 6 months and 12 months
  Impact of statin treatment(which will be given for 6 months) compared to no intervention or lifestyle modification on liver steatosis and fibrosis. Liver steatosis will be assessed by sonographic liver fat quantification (hepatorenal sonographic index.
change from baseline in liver fibrosis at 6 months | baseline, 6 months and 12 months
  Impact of statin treatment(which will be given for 6 months) compared to no intervention or lifestyle modification on liver fibrosis. Liver fibrosis will be assessed by Real-Time shear wave elastography.

SECONDARY OUTCOMES:
endothelial function in Non-Alcoholic Fatty Liver Disease (NAFLD) patients | 12 months
  measurement of endothelial function in NAFLD patients and finding the correlation between the degree of endothelial dysfunction and the severity of fatty liver disease. Endothelial function will be assessed by brachial artery flow-mediated (FMD) measurement at diagnosis and after 6 and 12 months. The severity of fatty liver disease will be assessed by liver elastography and sonographic liver fat quantification
relationship between blood parameters and liver steatosis and fibrosis | 12 months
  levels of liver enzymes, liver synthetic function, blood lipids, insulin resistance, ferritin, adiponectin, C reactive protein, Tumor necrosis factor alpha and ceruloplasmin and their correlation with liver steatosis and fibrosis
relationship between blood parameters and endothelial function | at diagnosis and after 6 months and 12 months
  levels of liver enzymes, liver synthetic function, blood lipids, insulin resistance, ferritin, adiponectin, C reactive protein, tumor necrosis factor alpha and ceruloplasmin and their correlation with endothelial function
change from baseline in endothelial function at 6 months | at diagnosis 6 months and 12 months
  Impact of statin treatment(which will be given for 6 months) compared to no intervention or lifestyle modification on endothelial function. Endothelial function will be assessed by flow mediated dilatation (FMD) of brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Ben-Ari, MD, Principal Investigator — Sheba Medical Center, Ramat Gan, Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel